CLINICAL TRIAL: NCT04196634
Title: Risk Assessment for Prolonged Sickness Absence Due to Musculoskeletal Conditions
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oslo Metropolitan University (Other)
Collaborators: Norwegian Labour and Welfare Administration (Other)
Responsible Party: Sponsor
Other Study IDs: NSD 861249
Record Dates: First submitted 2019-11-27; First posted 2019-12-12 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2022-08

CONDITIONS: Musculoskeletal Pain Disorder
Keywords: Risk Assessment
MeSH Terms: conditions — Collagen Diseases | interventions — Risk Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People on sick leave: People on sick leave due to musculoskeletal conditions for at least 4 weeks.
  Interventions: Other: Risk assessment

INTERVENTIONS:
Other: Risk assessment — People on sick leave due to musculoskeletal conditions will be screened for potential risk factors for prolonged sickness absence. No intervention will be given.

SUMMARY:
Musculoskeletal (MSK) conditions are a leading cause of years lived with disability worldwide and for the last decade they have also been the most common cause of sickness absence and disability pension in Norway.

Although most sickness absence is short-termed, a small proportion of people with MSK conditions are on long-term sick leave, contributing to large cost due to disbursement of benefits, productivity loss and extensive use of health care. There is growing evidence that long-term sickness absence is harmful to mental and physical health, with a reduced probability of return to work (RtW) with prolonged sickness absence. Thus, focusing on early RtW in people on sick leave due to MSK conditions is important to reduce the burden on both the individual and the society. However, to provide interventions to reduce the duration of sickness absence to all people on sick leave would require enormous resources. By targeting those at risk of long-term sickness absence, resources may be used differently, e.g. more resource-saving. By using information on modifiable risk factors from simple risk assessment tools, health care providers and other stakeholders may facilitate RtW in a better way.

The overall purposes of this project are 1) to identify the most accurate screening tool to identify people at a high risk of prolonged sickness absence due to a MSK condition, and 2) to investigate severity of MSK health, health-related quality-of-life, health care consumption, and costs across different risk profiles in people on sick leave due to MSK conditions. We will use registered data on sickness absence from 1 year before to 1 year after inclusion in the study.

DETAILED DESCRIPTION:
Main aims are:

* To compare the predictive ability of the STarT MSK tool and the ÖMPSQ-SF, and other established risk factors for long-term sickness absence (e.g. symptoms of depression and emotional distress, low motivation for returning to work, low self-efficacy, work expectancies) for identifying prolonged sickness absence at 6- and 12-months follow-up due to MSK conditions
* To develop a prognostic model to predict risk of prolonged sickness absence at 12-month follow-up in people with MSK conditions
* To assess predictors for high costs (productivity loss and health care use) at 6- and 12-months follow-up in people on sick leave due to MSK conditions

The study will also include additional methodological and descriptive aims.

Prior to the data collection we translated and culturally adapted the Keele STarT MSK and MSK-HQ following the Beaton guidelines.

The study is conducted within the Norwegian Welfare and Labor Administration (NAV) system in collaboration with OsloMet - Oslo Metropolitan University. Data on sickness absence from the NAV registry will be retrieved prospectively in the period from study inclusion to 12 months follow-up, and retrospectively 12 months prior to inclusion in the study.

Previous studies show that 30-40% of people with MSK conditions have not RtW after 3 to 12 months. In order to conduct analyses including 15- 20 predictor variables, we aim at including 500-600 people on sick leave due to MSK conditions. As the main outcomes are collected through registries, we do not expect any dropouts.

ELIGIBILITY:
Inclusion Criteria:

* People older than 18 years on sick leave due to musculoskeletal pain for at least 4 weeks

Exclusion Criteria:

* People on sick leave for other pain conditions or diseases
* People not able to read or write Norwegian or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female gender is a risk factor for developing musculoskeletal conditions, so we expect more women to be included in the study.
Study Population: People on sick leave due to musculoskeletal pain conditions in Norway were invited to participate. Eligible participants had to log on to their personal sickness absence website at the Norwegian Welfare and Labor Administration to be able to see a link to the project.
Sampling Method: Non-Probability Sample
Enrollment: 560 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Sickness absence days | 12 months
  Total number of absence days during 12 months of follow-up adjusted for percentage of work and percentage of sickness absence. Register data from the national health and welfare services
Time to sustainable return to work | 12 months
  The time until full sustainable return to work, i.e. at least 4 weeks without relapse during 12 months of follow-up. Register data from the national health and welfare services
Probability of return to work | 12 months
  Probability of working (i.e. not receiving medical benefits) each month during 12 months of follow-up, measured as repeated events. Register data from the national health and welfare services
Proportion who have returned to work | 12 months
  Proportion of people with sustainable return to work (at least 4 weeks) at 12 months. Register data from the national health and welfare services
Health care costs | 12 months
  Use of health care will be collected from public registries including Norwegian Patient Registry (NPR), Municipal Patient and User Registry (KPR) and Control and Payment of Health Refunds (KUHR).
Sickness absence costs | 12 months
  Sickness absence costs will be calculated based on data from the NAV registry

SECONDARY OUTCOMES:
Musculoskeletal Health Questionnaire (MSK-HQ) | Baseline and 4 weeks
  14 questions scored on a 0-4-point scale, summed up to a 0 to 56 points score, with higher score indicating better musculoskeletal health.
EuroQol 5 Dimensions (EQ5D-5L) | Baseline and 4 weeks
  The EQ5D-5L covers five domains: mobility, self-care, activities of daily living, pain/discomfort, and anxiety/depression, scored on a 5-point scale from 0 (worst imaginable health) to 5 (best imaginable health). Responses can be transformed into an index ranging from -0.59 to 1, where -0.59 represents worst possible state and 1 represents perfect health. The EQ5D Visual Analogue Scale (VAS) is also included, which is a question asking about the respondent's self-rated health on a vertical 0 to 100 visual analog scale, with 100 being best health.
Institute of Medical Technology Assessment (iMTA) Productivity Cost Questionnaire (iPCQ) | Baseline and 4 weeks
  Measure and value health-related productivity loss for both paid and unpaid work. The instrument is found to be suitable for measuring absenteeism from paid work and productivity loss related to unpaid labor. Nine questions related to paid work and three questions related to unpaid work.
Sickness absence days | 6 months
  Total number of absence days during 6 months of follow-up adjusted for percentage of work and percentage of sickness absence. Register data from the national health and welfare services
Time to sustainable return to work | 6 months
  The time until full sustainable return to work, i.e. at least 4 weeks without relapse during 6 months of follow-up. Register data from the national health and welfare services
Proportion who have returned to work | 6 months
  Proportion of people with sustainable return to work (at least 4 weeks) at 6 months. Register data from the national health and welfare services
Probability of return to work | 6 months
  Probability of working (i.e. not receiving medical benefits) each month during 6 months of follow-up, measured as repeated events. Register data from the national health and welfare services
Health care costs | 6 months
  Use of health care will be collected from public registries including Norwegian Patient Registry (NPR), Municipal Patient and User Registry (KPR) and Control and Payment of Health Refunds (KUHR).
Sickness absence costs | 6 months
  Sickness absence costs will be calculated based on data from the NAV registry

OTHER OUTCOMES:
Keele STarT MSK Screening tool | Baseline and 4 weeks
  The STarT MSK consists of 10 items and the scores are summarized to a 0-12 score, with risk groups being categorized as follow: 0-4= low risk; 5-8= medium risk; 9-12= high risk of developing long-term pain or disability.
Örebro Musculoskeletal Pain Screening Questionnaire short form (ÖMPSQ -sf) | Baseline and 4 weeks
  ÖMPSQ-sf contains 10 questions that are summed up to 0 to 100 score, with higher score indicating higher risk developing work disability.
Work conflict | Baseline and 4 weeks
  Single question on work conflict: "Did you experience conflict(s) with your employer before you got sick-listed?" (Yes/No)
Work satisfaction | Baseline and 4 weeks
  Measured with a single question: "If you take into consideration your work routines, management, salary, promotion possibilities and work mates, how satisfied are you with your job?" Measured on a numeric rating scale, 0=Not satisfied at all, 10=Completely satisfied
  Measured with a single question: "Do you want to return to the same work/position or do you wish you had another work/position?" Answered with: Same work/position / Another work/position.
Work ability | Baseline and 4 weeks
  Measured with a single question from the Work Ability Index: "Assume that your work ability at its best has a value of 10 ponts. How many points would you give to your current work ability?" Measured on a numeric rating scale where 0 means that you cannot currently work at all, 10 means that your work ability is at its best right now.
Return to work expectancy | Baseline and 4 weeks
  Measured with a single question: "For how long do you believe you will be sick listed from today?" Answered with: Not at all / Less than 1 month / 1-2 months / 2-4 months / 4-10 months / More than 10 months
Demographic variables | Baseline
  Gender, age, diagnosis
Change in condition | 4 weeks
  7-point global rating of change: "Could you please state the amount of change concerning your musculoskeletal symptoms compared to when you first filled out this questionnaire". Answered with: Much better / Better / Slightly better / Unchanged / Slightly worse / Worse / Much worse

CONTACTS AND LOCATIONS:
Overall Officials: Margreth Grotle, Prof, Principal Investigator — Oslo Metropolitan University
Locations (1):
- Oslo Metropolitan University, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Killingmo RM, Tveter AT, Pripp AH, Tingulstad A, Maas E, Rysstad T, Grotle M. Modifiable prognostic factors of high societal costs among people on sick leave due to musculoskeletal disorders: findings from an occupational cohort study. BMJ Open. 2024 Mar 1;14(3):e080567. doi: 10.1136/bmjopen-2023-080567. PMID 38431296
- [Derived] Munk Killingmo R, Tveter AT, Smastuen MC, Storheim K, Grotle M. Comparison of self-reported and public registered absenteeism among people on long-term sick leave due to musculoskeletal disorders: criterion validity of the iMTA Productivity Cost Questionnaire. Eur J Health Econ. 2021 Aug;22(6):865-872. doi: 10.1007/s10198-021-01294-0. Epub 2021 Jun 1. PMID 34061299
- [Derived] Tveter AT, Oiestad BE, Rysstad TL, Aanesen F, Tingulstad A, Smastuen MC, Grotle M. Risk assessment for prolonged sickness absence due to musculoskeletal disorders: protocol for a prospective cohort study. BMC Musculoskelet Disord. 2020 May 25;21(1):326. doi: 10.1186/s12891-020-03354-7. PMID 32450820

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Statistical Analysis Plan - Prognostic factors (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/34/NCT04196634/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan - Prognostic model (2023-02-06): https://cdn.clinicaltrials.gov/large-docs/34/NCT04196634/SAP_001.pdf